CLINICAL TRIAL: NCT04499950
Title: A Phase II Single Arm Adaptive Weight Loss Study in Women With Early Stage Breast Cancer
Brief Title: Adaptive Nutrition and Exercise Weight Loss (A-NEW) Study
Acronym: A-NEW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: American Institute for Cancer Research (Other); Breast Cancer Research Foundation (Other); Hopkins-WellSpan Cancer Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: IRB00223131
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Overweight or Obesity
MeSH Terms: conditions — Breast Neoplasms; Overweight; Obesity | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination; Naltrexone; Bupropion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SLOW-BWL (Experimental): All patients will receive the POWER-remote behavioral weight loss intervention (BWL) and have a behavioral coach for the duration of the 6 month study. During months 1-3, the behavioral coach will call weekly. From months 4-6, the behavioral coach will call monthly. At week 9, those who lose <5%, designated slow responders, will continue BWL and initiate Contrave (SLOW-BWL). The SLOW-BWL arm will receive at least 16 weeks of Contrave [as per the Food and Drug Administration (FDA) recommended administration] starting at week 9 and discontinue if ≥5% weight loss is not achieved at month 6.
  Interventions: Drug: Contrave; Behavioral: Behavioral Weight Loss
- FAST-BWL (Active Comparator): All patients will receive the POWER-remote behavioral weight loss intervention (BWL) and have a behavioral coach for the duration of the 6 month study. During months 1-3, the behavioral coach will call weekly. From months 4-6, the behavioral coach will call monthly. At week 9, those who lose ≥5%, designated fast responders, will continue with BWL alone (FAST-BWL)
  Interventions: Behavioral: Behavioral Weight Loss

INTERVENTIONS:
Drug: Contrave — Initiate Contrave at 1 tab in morning (AM) for Week 9; then 1 tab in AM and 1 tab in evening (PM) for Week 10; then 2 tab in AM and 1 tab in PM for Week 11; then 2 tab in AM and 2 tab in PM for week 12; then constant dose for months 4-6.
  Other Names: Naltrexone/Bupropion
  Arms: SLOW-BWL
Behavioral: Behavioral Weight Loss — 6 months of behavioral weight loss. First 3 months are weekly calls with coach and then transition to monthly calls for months 4-6.

SUMMARY:
This is a single arm phase II study designed to determine the effects of pharmacotherapy and a remote behavioral weight loss intervention on weight loss in breast cancer survivors who are overweight or obese, and the impact of successful weight loss on serum biomarkers and gut microbiome.

DETAILED DESCRIPTION:
The investigators will evaluate the extent to which implementation of a chronic weight loss medication, Contrave® (Naltrexone/Bupropion), is associated with achieving ≥5% weight loss. All patients will receive the POWER-remote behavioral weight loss intervention (BWL) and have a behavioral coach for the duration of the 6 month study. During months 1-3, the behavioral coach will call weekly. From months 4-6, the behavioral coach will call monthly. At week 9, those who lose ≥5%, designated fast responders, will continue with BWL alone (FAST-BWL) while those who lose <5%, designated slow responders, will continue BWL and initiate Contrave (SLOW-BWL). The SLOW-BWL arm will receive at least 16 weeks of Contrave (as per Federal Drug Administration [FDA] recommended administration) starting at week 9 and discontinue if ≥5% weight loss is not achieved at month 6. During month 3, all participants continue to have weekly calls with the behavioral coach and will be asked about symptoms, which may be related to initiation of pharmacotherapy; any symptoms are reported to the PI for further evaluation. In addition to total weight loss, the investigators will evaluate biomarkers associated with obesity, microbiome and cardiometabolic factors.

ELIGIBILITY:
Inclusion Criteria:

* Female, at least 3 months after completion of local therapy (e.g. surgery, radiation), and if applicable, adjuvant chemotherapy
* Diagnosed within 10 years with histologically-confirmed ductal carcinoma in situ (DCIS) or stage I-III invasive carcinoma of the breast
* Up to date with recommended screening mammography within one year
* Current BMI ≥ 30 kg/m2 or BMI 27.0-29.9 kg/m2 with hypertension, non-insulin dependent diabetes or hyperlipidemia; and weight ≤ 400 lbs
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Willingness to change diet, physical activity, track behaviors, engage in weekly and monthly contacts and visit, and take chronic weight loss medication
* Able to read and write the English language without assistance and daily access to the e-mail and/or smartphone
* Patient is aware of her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Serious/uncontrolled medical condition at the discretion of the Protocol Chair/designee likely to hinder accurate measurement of weight or any condition for which weight loss is contraindicated or would affect adipokine and inflammatory markers (e.g. active malignancy, end stage renal disease on dialysis, cirrhosis, autoimmune disease, adrenal disease, uncontrolled hypertension, seizure disorder, and history of bariatric surgery)
* Pregnant or nursing within past 6 months, or plans to become pregnant in the next year
* Currently enrolled or planning to enroll in a weight loss program (e.g. Weight Watchers, Jenny Craig, Nutrisystem and Medifast) or to take a chronic weight loss medication.
* Diabetes on insulin or sulfonylureas within the past 3 months
* Unstable psychiatric disorder or bulimia/anorexia nervosa
* Alcohol, nicotine or substance abuse; or undergoing abrupt discontinuation of alcohol, benzodiazepine, barbiturate or anti-epileptic drug
* Use of the following medications are excluded:

  * Monoamine oxidase (MAO) inhibitors (must be >14 days from discontinuation)
  * Thyroid medication use unless on stable doses for at least the past 3 months
  * Buproprion containing products or opiate agonists (must be >14 days from discontinuation)
  * Medications that cause weight loss (e.g., lorcaserin, phentermine, orlistat, Qsymia, Contrave) within the past 3 months
  * Medications that are likely to cause weight gain or prevent weight loss (e.g., corticosteroids, lithium, olanzapine, risperidone, clozapine, oral contraceptive pills, hormone replacement therapy) within the past 3 months. NOTE: An exception to this is that SSRI's and SNRI's are allowed if participant has been on stable doses for at least 3 months (if discontinued, a washout of 2 weeks from prior selective serotonin reuptake inhibitor (SSRI)/Serotonin-norepinephrine reuptake inhibitor (SNRI) use is required).
  * Medications that may affect adipokine or inflammatory markers (e.g., metformin, glitazones, steroids, angiotensin converting enzyme (ACE) inhibitors, beta blockers and statins) unless on stable doses ≥3 months prior to registration (if discontinued, a washout of 2 weeks from prior use is required). Concurrent NSAIDs are allowed if use is limited to <3 times per week; chronic NSAIDs are permitted on study only if use has been ≥3 times per week for at least 3 months prior to registration and is expected to continue.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sheng, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SLOW-BWL | FAST-BWL
Started | 38 | 15
Completed | 38 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SLOW-BWL | FAST-BWL | Total
Number analyzed (Participants) | 38 | 15 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 10 | 42
  >=65 years | 6 | 5 | 11
Age, Continuous [Median (Full Range); unit: years] | 56.5 [30 to 73] | 61 [40 to 73] | 59 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 15 | 53
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/ Caucasian | 24 | 13 | 37
  Black or African American | 12 | 1 | 13
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 15 | 53
Breast Cancer Stage [Count of Participants; unit: Participants] — Breast cancer stage at study entry: Ductal carcinoma in situ (DCIS), Stage 1, Stage 2 or Stage 3.
  Staging done with The American Joint Committee on Cancer (AJCCC) Version 8. Higher stage is worse.
  Participants
    Stage 0 (Ductal carcinoma in situ (DCIS)) | 2 | 3 | 5
    Stage 1 | 23 | 6 | 29
    Stage 2 | 8 | 2 | 10
    Stage 3 | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With 5 Percent Weight Loss (in SLOW-BWL)
Description: To assess the rate of SLOW-BWL patients attaining at least 5% weight loss of their baseline body weight at 6 months with the addition of Contrave to BWL at week 9.
Time Frame: 6 months
Population: Only 32 participants in the SLOW-BWL arm completed intervention per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | SLOW-BWL
Number analyzed (Participants) | 32
Participants | 16

2. Secondary Outcome: Change in Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function - Short Form Questionnaire Among FAST-BWL vs SLOW-BWL, as Well as Participants Who Achieve ≥5% Weight Loss at 6 Months vs Those Who Are Unable to
Description: To report the change in scores at 2 and 6 months to baseline among FAST-BWL vs SLOW-BWL arms for Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function. The total score ranges from 33.5 to 61.7. The higher the score, the better the physical function.
Time Frame: Baseline, 2 months and 6 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | SLOW-BWL | FAST-BWL
Number analyzed (Participants) | 38 | 15
units on a scale
  Baseline to 2 months | 2 [0 to 5] | 3 [-2 to 6]
  2 months to 6 months | 0.0 [-0.8 to 3.3] | 1.1 [0.0 to 9.0]

3. Secondary Outcome: Change in Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference - Short Form Questionnaire Among FAST-BWL vs SLOW-BWL, as Well as Participants Who Achieve ≥5% Weight Loss at 6 Months vs Those Who Are Unable to
Description: To report the change in scores at 2 and 6 months to baseline among FAST-BWL vs SLOW-BWL arms for Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference. The total score ranges from 41.0-67.4. The lower the score, the better the pain interference.
Time Frame: Baseline, 2 months and 6 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | SLOW-BWL | FAST-BWL
Number analyzed (Participants) | 38 | 15
units on a scale
  Baseline to 2 months | -1.1 [-4.1 to 1.3] | 0.0 [-7.2 to 0.0]
  2 months to 6 months | 0.0 [-1.3 to 1.3] | 0.0 [-4.2 to 0.0]

4. Secondary Outcome: Change in Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue - Short Form Questionnaire Among FAST-BWL vs SLOW-BWL, as Well as Participants Who Achieve ≥5% Weight Loss at 6 Months vs Those Who Are Unable to
Description: To report the change in scores at 2 and 6 months to baseline among FAST-BWL vs SLOW-BWL arms for Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue. The total score ranges from 39.6 to 62.0. The lower the score, the less the fatigue.
Time Frame: Baseline, 2 months and 6 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- SLOW-BWL Baseline - 2 Months: All patients will receive the POWER-remote behavioral weight loss intervention (BWL) and have a behavioral coach for the duration of the 6 month study. During months 1-3, the behavioral coach will call weekly. From months 4-6, the behavioral coach will call monthly. At week 9, those who lose <5%, designated slow responders, will continue BWL and initiate Contrave (SLOW-BWL). The SLOW-BWL arm will receive at least 16 weeks of Contrave [as per the Food and Drug Administration (FDA) recommended administration] starting at week 9 and discontinue if ≥5% weight loss is not achieved at month 6.
  Contrave: Initiate Contrave at 1 tab in morning (AM) for Week 9; then 1 tab in AM and 1 tab in evening (PM) for Week 10; then 2 tab in AM and 1 tab in PM for Week 11; then 2 tab in AM and 2 tab in PM for week 12; then constant dose for months 4-6.
  Behavioral Weight Loss: 6 months of behavioral weight loss. First 3 months are weekly calls with coach and then transition to monthly calls for months 4-6.
- FAST-BWL Baseline - 2 Months: All patients will receive the POWER-remote behavioral weight loss intervention (BWL) and have a behavioral coach for the duration of the 6 month study. During months 1-3, the behavioral coach will call weekly. From months 4-6, the behavioral coach will call monthly. At week 9, those who lose ≥5%, designated fast responders, will continue with BWL alone (FAST-BWL)
  Behavioral Weight Loss: 6 months of behavioral weight loss. First 3 months are weekly calls with coach and then transition to monthly calls for months 4-6.
Arm/Group | SLOW-BWL Baseline - 2 Months | FAST-BWL Baseline - 2 Months
Number analyzed (Participants) | 38 | 15
units on a scale
  Baseline to 2 months | 0.0 [-5.0 to 3.2] | 0.0 [-4.1 to 3.9]
  2 months to 6 months | 1.6 [-2.0 to 5.3] | -0.7 [-3.4 to 3.1]

5. Secondary Outcome: Change in Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Depression - Among FAST-BWL vs SLOW-BWL, as Well as Participants Who Achieve ≥5% Weight Loss at 6 Months vs Those Who Are Unable to
Description: To report the change in scores at 2 and 6 months to baseline among FAST-BWL vs SLOW-BWL arms for Patient-Reported Outcomes Measurement Information System (PROMIS) Depression. The total score ranges from 37.1-71.4. The lower the score, the less depression.
Time Frame: Baseline, 2 months and 6 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | SLOW-BWL | FAST-BWL
Number analyzed (Participants) | 38 | 15
units on a scale
  Baseline to 2 months | 0.0 [-6.20 to 0.0] | 0.0 [-1.50 to 0.80]
  2 months to 6 months | 0.0 [-2.0 to 0.0] | -1.8 [-8.4 to 0.0]

6. Secondary Outcome: Change in Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety - Among FAST-BWL vs SLOW-BWL, as Well as Participants Who Achieve ≥5% Weight Loss at 6 Months vs Those Who Are Unable to
Description: To report the change in scores at 2 and 6 months to baseline among FAST-BWL vs SLOW-BWL arms for Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety. Scores range 36.3-71.5, with higher scores representing more severe anxiety symptoms.
Time Frame: Baseline, 2 months and 6 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | SLOW-BWL | FAST-BWL
Number analyzed (Participants) | 38 | 15
units on a scale
  Baseline to 2 months | 0.0 [-3.7 to 1.3] | 0.0 [-0.6 to 2.4]
  2 months to 6 months | 0 [-6 to 2] | -1 [-3 to 1]

7. Secondary Outcome: Change in Scores on the Medical Outcomes Study (MOS) Sexual Functioning Scale Among FAST-BWL vs SLOW-BWL, as Well as Participants Who Achieve ≥5% Weight Loss at 6 Months vs Those Who Are Unable to
Description: To report the change in scores at 2 and 6 months to baseline among FAST-BWL vs SLOW-BWL arms for Medical Outcomes Study (MOS) Sexual Function. Score range 0-100 with higher score indicating less functioning.
  Four items are rated on a 5-point scale (1=not a problem, 2=little of a problem, 3=somewhat of a problem, 4=very much of a problem, and 5=not applicable).
Time Frame: Baseline, 2 months and 6 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | SLOW-BWL | FAST-BWL
Number analyzed (Participants) | 38 | 15
units on a scale
  Baseline to 2 months | 0 [-9 to 0] | 0 [-12 to 0]
  2 months to 6 months | 0 [0 to 0] | 0 [-12 to 0]

8. Secondary Outcome: Change in Scores on Functional Assessment of Cancer Therapy-Endocrine Subscale (FACT-ES) Among FAST-BWL vs SLOW-BWL, as Well as Participants Who Achieve ≥5% Weight Loss at 6 Months vs Those Who Are Unable to
Description: To report the change in scores at 2 and 6 months to baseline among FAST-BWL vs SLOW-BWL arms for Functional Assessment of Cancer Therapy-Endocrine Subscale (FACT-ES). Scores ranging from 39.0 to 73.0. Higher scores indicate greater impact from symptoms.
Time Frame: Baseline, 2 months and 6 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | SLOW-BWL | FAST-BWL
Number analyzed (Participants) | 38 | 15
units on a scale
  Baseline to 2 months | 3 [-2 to 6] | 2 [1 to 4]
  2 months to 6 months | 6 [0 to 10] | 4 [2 to 8]

9. Other Pre Specified Outcome: Number of Patients With 5% Weight Loss (in FAST-BWL)
Description: To assess the proportion of women in the FAST-BWL arm who maintain ≥5% weight loss at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | FAST-BWL
Number analyzed (Participants) | 15
Participants | 13

ADVERSE EVENTS:
Time Frame: Initiation of drug up to 6 months
Arm/Group | SLOW-BWL | FAST-BWL
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/15
Other Adverse Events (participants affected / at risk) | 28/38 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SLOW-BWL (N=38) | FAST-BWL (N=15)
constipation (Gastrointestinal disorders) | 20 | 2
Nausea (Gastrointestinal disorders) | 16 | 1
dry mouth (Gastrointestinal disorders) | 14 | 1
Diarrhea (Gastrointestinal disorders) | 10 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 1
Bloating (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 12 | 0
Anxiety (Psychiatric disorders) | 6 | 0
Headache (Nervous system disorders) | 9 | 0
Dizziness (Nervous system disorders) | 3 | 1
Fatigue (General disorders) | 8 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hot flashes (Vascular disorders) | 5 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Tremor (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04499950/Prot_SAP_000.pdf